CLINICAL TRIAL: NCT06917131
Title: Royal Jelly as a Strategy to Modulate Inflammation and Oxidative Stress in Patients With Systemic Arterial Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Denise Mafra21
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Cardiovascular Diseases (CVD); Inflammation
Keywords: royal jelly; inflammation; Hypertension; cardiovascular diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Inflammation | interventions — royal jelly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Royal Jelly Group (Experimental): Participants will receive 2 capsules per day, providing the dosage of 300mg of royal jelly for 2 months (8 weeks).
  Interventions: Dietary Supplement: Royal Jelly
- Placebo Group (Placebo Comparator): The placebo group will receive 2 capsules per day (containing microcrystalline cellulose and magnesium stearate in colored gelatin capsules capable of masking the appearance of the internal content), at the same time for 2 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Royal Jelly — Participants will receive 2 capsules per day, providing the dosage of 300mg of royal jelly for 2 months (8 weeks).
  Arms: Royal Jelly Group
Dietary Supplement: Placebo — The placebo group will receive 2 capsules per day (containing microcrystalline cellulose and magnesium stearate in colored gelatin capsules capable of masking the appearance of the internal content), at the same time for 2 months.
  Arms: Placebo Group

SUMMARY:
The study aims to evaluate the effect of the royal jelly on inflammation and oxidative stress in participants with systemic arterial hypertension. A longitudinal double-blind randomized clinical trial will be carried out, involving hypertensive participants for two months.

DETAILED DESCRIPTION:
Royal jelly (RG) is considered a superfood that has been used in traditional medicine and dietary supplementation due to its antioxidant, anti-inflammatory, immunomodulatory, and regenerative properties. The antioxidant and anti-inflammatory effects of GR highlight its potential as a natural supplement for the prevention and management of several health conditions. Although in vitro and animal model data are promising, clinical studies are still needed to validate the effects of royal jelly in human populations.

ELIGIBILITY:
Inclusion Criteria:

* patients using one to three antihypertensive medications, undergoing regular follow-up at the HUAP Medical Clinic for more than 6 months and without the need for changes in medication doses in the last 3 months.

Exclusion Criteria:

* Patients with autoimmune and infectious diseases, diabetes, chronic kidney disease, liver disease, cancer and AIDS will be excluded; pregnant women; those using catabolic drugs or antibiotics; use of antioxidant vitamin supplements, prebiotics, probiotics, symbiotics, habitual intake of royal jelly, and who are allergic to cornstarch or report having an allergy to bee stings will also be excluded. Patients with acute myocardial infarction (AMI) and/or stroke (CVA) in the last 6 months will also be excluded; with HAS stages 2 or 3.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change of inflammatory status in the participants | Baseline and 8 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory and oxidative stress biomarkers: NfkB, Nrf2, interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-alpha), C-reactive protein (CRP), antioxidant enzymes.

CONTACTS AND LOCATIONS:
Overall Officials: Ludmila Cardozo, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
Participant data will not be public to other research unless necessary.